CLINICAL TRIAL: NCT01124877
Title: 26 Week Open Label Extension Study Evaluating The Safety And Tolerability Of Flexible Doses Of Oral Ziprasidone In Children And Adolescents With Bipolar I Disorder (Manic Or Mixed)
Brief Title: Safety And Tolerability Of Flexible Doses Of Oral Ziprasidone In Children And Adolescents With Bipolar I Disorder (Manic Or Mixed)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1281197
Record Dates: First submitted 2010-05-14; First posted 2010-05-17 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Bipolar Disorder
Keywords: Children and Adolescents with Bipolar I Disorder (manic or mixed)
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open (Other)
  Interventions: Drug: ziprasidone oral capsules

INTERVENTIONS:
Drug: ziprasidone oral capsules — Oral ziprasidone capsules of 20 mg, 40 mg, 60 mg, and 80 mg strength will be provided. Subjects will be dosed daily for 26 weeks using a flexible dose design with a minimal dose range of 40mg twice a day (BID) to a maximum dose range of 80 mg BID. For subjects weighing <45 kg, the doses will range from 20 mg BID to 40 mg BID.
  Other Names: Zeldox, Geodon

SUMMARY:
The purpose of this study is to assess the safety and tolerability of ziprasidone during a long-term open label study in children and adolescents (ages 10-17) with Bipolar I Disorder (Manic or Mixed).

ELIGIBILITY:
Inclusion Criteria:

* The subjects must have received study medication in Study A1281196.
* In the investigator's opinion, the subject must be likely to continue to benefit from antipsychotic therapy and must have been free from any clinically significant safety concerns during the preceding double blind study.

Exclusion Criteria:

* Subjects who require treatment with drugs that are known to consistently prolong the QT interval.
* Subjects who are judged by the investigator as being at imminent risk of suicide.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in blood pressure and pulse Change from baseline in electrocardiogram (QTc) Change from Baseline in Clinical Global Impression of Severity Scale (CGI-S) | weeks 1, 2, 6, 10, 14, 18, 22, and 26
Change from baseline in Physical exam | week 26
Change from baseline in Clinical laboratory tests | weeks 2, 6, 18,26
Change from baseline in body weight, height, BMI, BMI z score, and waist circumference | weeks 6, 26
Adverse events -Only number of subjects with adverse events or serious adverse events Columbia Suicide Severity Rating Scale Change from Baseline in Child Depression Rating Scale - Revised (CDRS-R) | weeks 1, 2, 6, 10, 14, 18, 22, and 26

SECONDARY OUTCOMES:
Change from Baseline in Young Mania Rating Scale (YMRS) | weeks 2, 6, 18, and 26
Change from Baseline in Children's Problem Behavior and Aggression Questionnaire (CPBAQ) | weeks 2, 6, 18, and 26
Change from Baseline in Child Health Questionnaire | weeks 6 and 26
Change from Baseline in School Placement Questionnaire | weeks 6 and 26
Change from Baseline in CNS Vital Signs Cognitive Test Battery | weeks 6 and 26
Change from Baseline in CNS Vital Signs Cognitive Test Sedation Item | weeks 6 and 26
Change from Baseline in Simpson-Angus Rating Scale (SARS) | weeks 1, 2, 6, 10, 14, 18, 22 and 26
Change from Baseline in Barnes Akathisia Rating Scale (BAS) | weeks 1, 2, 6, 10, 14, 18, 22 and 26
Change from Baseline in Abnormal Involuntary Movement Scale (AIMS) | weeks 1, 2, 6, 10, 14, 18, 22 and 26
Change from Baseline in Childrens Global Assessment Scales | weeks 2, 6, 18, and 26
Change from Baseline in Tanner Adolescent Pubertal Self-Assessment | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281197&StudyName=Safety%20And%20Tolerability%20Of%20Flexible%20Doses%20Of%20Oral%20Ziprasidone%20In%20Children%20And%20Adolescents%20With%20Bipolar%20I%20Disorder%20%28Manic%20Or%20Mixed%29